CLINICAL TRIAL: NCT03597841
Title: Turkish Prospective Cohort Study on Carbapenem Resistant Klebsiella Pneumonia Bacteremia: a National Multicenter Observational Study
Brief Title: Turkish Prospective Cohort Study on Carbapenem Resistant Klebsiella Pneumonia Bacteremia
Acronym: THREAT
Status: Completed | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Burcu Isler, Coordinator, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2018.151.IRB1.018
Record Dates: First submitted 2018-07-09; First posted 2018-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Klebsiella Pneumonia; Bacteremia
Keywords: Monotherapy; Combination therapy; Colistin-resistant; Klebsiella Pneumonia; Bacteremia; Blood stream infection
MeSH Terms: conditions — Bacteremia | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with CRKp BSI:Combination therapy
  Interventions: Drug: Combination therapy
- Patients with CRKp BSI: Monotherapy

INTERVENTIONS:
Drug: Combination therapy — Patients who are given combination therapy will be allocated to this group.
  Groups: Patients with CRKp BSI:Combination therapy

SUMMARY:
Carbapenem-resistant Klebsiella pneumonia (CRKp) blood stream infections (BSI) cause substantial mortality among hospitalized patients. Treatment options for CRKp infections are limited and increasing resistance rates to few available drugs, i.e., colistin, is a big concern. This prospective multicenter observational study is designed to describe clinical characteristics and outcomes of patients with CRKp bacteremia in an oxacillinase-48 (OXA-48) endemic country to define predictors of mortality with a focus on the impact of mono versus combination therapies on mortality. The study will also investigate risk factors associated with colistin-resistant CRKp BSI.

DETAILED DESCRIPTION:
OBJECTIVES

MAIN OBJECTIVE

1. To compare the impact of combination therapy and monotherapy on mortality for patients with CRKp BSI

   SECONDARY OBJECTIVES
2. To identify predictors of mortality for patients with CRKp BSI
3. To compare the impact of appropriate and inappropriate empiric and targeted therapies on mortality for patients with CRKp BSI
4. To identify the risk factors for colistin resistance among patients with ColR CRKp BSI.

HYPOTHESES

MAIN HYPOTHESIS

1. Combination therapy is better than monotherapy to prevent 30-day mortality.

   i.Combination of one active drug with one inactive drug is not associated with lower probability of mortality as compared to monotherapy with one active drug if:
   * the inactive drug is carbapenem with a minimum inhibitory concentration (MIC) of ≥16 mg/L or
   * the inactive drug is any other antibiotic other than carbapenem or
   * the patient is in low mortality score

   ii.Combination of two or more active drugs is associated with lower probability of mortality as compared to monotherapy with one active drug.

   iii.For colistin resistant CRKp, monotherapy with one active drug is associated with lower probability of mortality as compared to combination therapies including carbapenem with a MIC of ≥16 mg/L or colistin.

   SECONDARY HYPOTHESES
2. Severe disease at BSI onset (admission to ICU, septic shock, INCREMENT-CPE (carbapenemase-producing Enterobacteriaceae) score 8-15, higher sequential organ failure assessment (SOFA) and Pitt bacteremia scores, Charlson Comorbidity Index ≥2, higher procalcitonin levels), carbapenemase type and carbapenem MIC of the isolate (CRKp isolates with a carbapenem MIC ≥16 mg/L, OXA-48 producing isolates), sequence type of the isolate (ST101 and ST258), colistin resistance delayed source control (>48 hours) and infection sources other than urinary tract are independent predictors of mortality.
3. Appropriate empirical therapy, early targeted therapy, are independent predictors of survival. For colistin susceptible CRKp, empirical use of colistin within 24 hours of BSI onset is associated with lower probability of mortality.
4. Previous colistin therapy, previous CRKp infection, previous intensive care unit (ICU) stay (last three months), length of hospital stay until index date is associated with colistin resistance. Mortality rates and length of hospital stay are higher among colistin resistant strains as compared to colistin susceptible strains.
5. Effect of treatment type on mortality is modified by disease severity.

STUDY DESIGN

Prospective cohort study.

Setting and study period

Fourteen tertiary care hospitals from the four most populous cities in Turkey (Istanbul, Ankara, Izmir, Bursa) are included in the study. Study period is scheduled to be 25 June 2018- 25 June 2019 or longer until pre-defined sample size is reached. Local investigators (infectious disease physicians and clinical microbiologists) will collect microbiological and clinical data. Site investigators will screen the microbiology laboratory logs daily to identify patients with CRKp bacteremia. All consecutive patients with CRKp bacteremia will be eligible to be evaluated for inclusion in the study. Patients who meet the inclusion criteria will be selected for the prospective cohort study and/or case-control study depending on colistin resistance pattern of the isolate. Site investigators will access patients' medical records and register relevant information using a web-based data entry system. Site investigators will also collect CRKp isolates and keep them in appropriate conditions until time of transfer for analysis. All CRKp isolates will be sent to the central microbiology laboratory for molecular analysis and colistin and ceftazidime-avibactam sensitivity testing.

Sample size

The expected mortality rate for CRKp BSI is approximately 40% based on previous studies (7, 12) To detect a 17% decrease in mortality rate with combination therapy as compared to monotherapy, we calculated an overall sample size of 178 (α=0.05, power=0.8) (STATA 15.0, power analysis for the cox proportional hazards model) (7). Considering withdrawals and incomplete data, we aimed to recruit 200 patients.

Given that we were able to recruit patients faster than expected within our study period (25 June 2018- 25 June 2019), we decided to increase our power to 0.9.

Follow up

Patients will be evaluated for microbiologic eradication on day 3 by control blood cultures and primary source cultures. If CRKp is not eradicated on day 3, consecutive cultures will be taken on day 7 and 14, as required. Patients will also be evaluated for clinical response on day 7 and day 14 using 7th and 14th day SOFA scores, C-reactive protein, procalcitonin and leucocyte levels and clinical signs of infection. All patients will be followed for 30 days after index date. If the patient is discharged before completion of the 30 days, he/she will be contacted by phone on day 30 to assess the outcome.

DEFINITIONS

CRKp: K. pneumonia non-susceptible to at least one carbapenem according to EUCAST 2018 breakpoints.

Colistin-resistant (ColR) CRKp: CRKp resistant to colistin according to EUCAST breakpoints

CRKp bacteremia: Presence of at least one set of blood culture positive for CRKp

CRKp BSI: Presence of at least one set of blood culture positive for CRKp with evidence of systemic inflammatory response.

Index date: The day of collection of the CRKp positive blood culture, infection onset, day 0.

Active drug: Antibiotic with in vitro activity against the CRKp isolate (antibiotic which the isolate is susceptible or intermediate to)

Inactive drug: Antibiotic without in vitro activity against the CRKp isolate (antibiotic which the isolate is resistant to)

Empiric therapy: Treatment administered following blood culture collection and prior to antimicrobial susceptibility test results

Targeted therapy: Treatment initiated or maintained after obtaining antimicrobial susceptibility test results

Appropriate therapy: Treatment regimen that includes at least one active drug initiated within 5 days of the index date and administered for at least 48 hours (24 hours for the patients who died within 2 days of the index date)

Early appropriate therapy: Treatment regimen that includes at least one active drug initiated within 2 days of the index date and administered for at least 48 hours (24 hours for the patients who died within 2 days of the index date)

Inappropriate therapy: Treatment regimen that does not include any active drugs and/or treatment administered for less than 48 h and/or treatment initiated after 5 days of the index date.

Monotherapy: Treatment with one active drug

Combination therapy: Treatment with more than one active drug

Primary bacteremia: Catheter-related bacteremia and bacteremia of unknown source

Secondary bacteremia: Identical CRKp growth from a specific body site within BSI window period (3 days before and 3 days after positive blood culture)

Polymicrobial bacteremia: Polymicrobial episodes (defined as ≥2 isolates of different microorganisms in samples taken ≤2 day apart from the same patient

Suspected source: The source of bacteremia determined by the attending physician according to the clinical presentation of the patient, rather than by the culture growth.

Source control: Central line removal, debridement, percutaneous or surgical drainage that are performed within 48 hours of BSI onset.

VARIABLES

Host variables: Age, sex, ward (ICU or non-ICU), hospital type and ward if transferred from another hospital, underlying diseases (Charlson Comorbidity Index), risk factors for acquisition of CRKp (previous infection: prior positive culture with CRKp, hospital stay for >48 hours in last three months, ICU stay for >48 hours in last three months, major surgery in previous month, antibiotic use in last three months: Carbapenem, colistin, other, invasive procedures performed within one week of BSI onset (insertion of central venous catheters, nasogastric tubes, foley catheters; endoscopy; endoscopic retrograde cholangiopancreatography; bronchoscopy; parenteral nutrition; mechanical ventilation), disease severity at index date: SOFA score, Pitt bacteremia score, INCREMENT-CPE score, presentation with septic shock, length of hospital stay until index date

Infection variables: Infection acquisition (Community-acquired vs. hospital-acquired), primary or secondary bacteremia, source control, procalcitonin & C-reactive protein & leucocyte at day 0, 7 and 14, creatinine and glomerular filtration rate (GFR).

Treatment variables: Antimicrobial therapy (duration, dosage (loading and maintenance), presence of prolonged infusion (only for carbapenems))

Microbiological variables: Automated system used for isolate identification and antimicrobial susceptibility testing in the local laboratory, susceptibility profile of the CRKp isolates, MICs for carbapenem, colistin, tigecycline and ceftazidime-avibactam, carbapenemase type, sequence type

MICROBIOLOGICAL STUDIES

Identification and antimicrobial susceptibility testing of CRKp isolates will be performed at local laboratories. MICs will be interpreted according to EUCAST (European Committee on Antimicrobial Susceptibility Testing) criteria. Colistin susceptibility test results will be confirmed and ceftazidime-avibactam susceptibility results will be determined at reference laboratory by broth microdilution. Molecular studies to identify carbapenem resistance genes, colistin resistance mechanisms and CRKp sequence types will be performed at the reference laboratory. Genetic relatedness of the isolates will also be determined at reference laboratory.

STATISTICAL ANALYSIS

Survivor and non-survivor patients with CRKp bacteremia will be compared to identify predictors of mortality. Continuous variables will be compared using t-tests or Mann-Whitney U tests. Categorical variables will be evaluated with the χ2 or Fisher's exact test. Two-tailed tests will be used to determine statistical significance and a p value of < 0.05 will be considered significant.

Effect of treatment type (mono vs. combination therapies, appropriate vs. inappropriate and early vs. late start empiric and targeted therapies) on clinical or microbiological response at day 7 (and 14 if applicable) and on mortality at day 30 will be assessed by logistic regression and cox proportional hazards model, respectively. Independent variables that are either identified from univariate analysis as statistically significant or reported in the literature as being associated with the outcome will be used as covariates. Interaction between treatment type and disease severity/mortality scores will also be assessed and stratified analyses according to disease severity will be performed. Survival curves will be obtained by Kaplan-Meier method and compared using log-rank test.

Propensity score for receiving combination therapy will be calculated using a logistic regression model. Age, sex, hospital, transfer from another hospital, history of hospitalization and antibiotic use, Charlson comorbidity index, ICU stay, SOFA score, Pitt bacteremia score, septic shock, procalcitonin level, infection acquisition type, source of infection will be included as independent variables in the model.

ColR CRKp cases will be compared with colistin-sensitive (ColS) controls in a nested case-control analysis. Competing risks of death for ColR CRKp BSI will be assessed.

Discriminating ability of the models will be assessed by estimating areas under the receiver operating characteristic (ROC) curves. Collinearity will be assessed by calculating variance inflation factors (VIFs) for each dependent variable in the analysis. Akaike information criteria (AIC) will be used for model selection.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥18 years old) with clinically significant CRKp bacteremia

Exclusion Criteria:

* Polymicrobial infection (except coagulase-negative staphylococci or other skin contaminants isolated from one blood culture bottle, which is considered contamination)
* Subsequent CRKp bacteremia episodes from the same patient

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult hospitalized patients (≥18 years old) with clinically significant CRKp bacteremia
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
30-day crude mortality | 1 month
  Death by any cause

SECONDARY OUTCOMES:
In-hospital mortality | 1 month
  Death by any cause during hospitalization
Clinical response at day 7 and 14 | day 7 and 14
  * Complete response: Improvement in clinical response resulting in ceasing of antibiotic therapy.
  * Partial response: Improvement in clinical response with continuation of antibiotic therapy.
  * No response: No improvement
Microbiologic eradication | day 3, 7 and/or 14
  * Established: No growth in follow-up cultures on day 3, 7 or 14
  * Presumed: No follow up cultures performed but clinical response is observed
  * Unknown: No follow up cultures performed, and no clinical response observed
Infection related mortality | 1 month
  Mortality attributed to the infection by the local investigators.
  * Attributable (directly related)
  * Contributable (indirectly related)
  * Non-related
Duration of hospital stay after infection | 1 month
  Duration of hospital stay after infection until day 30
ICU stay after infection | 1 month
  Duration of ICU stay after infection until day 30
Duration of antibiotic treatment | 1 month
  Total duration of antibiotic treatment
Recurrence | 1 month
  Recurrence of CRKp bacteremia within 30 days after clinical and/or microbiological response
Superinfection | 1 month
  Occurrence of any infection by a different organism during the 30-day period after the initial blood culture positive for CRKp.
Colistin resistance development | 1 month
  Isolation of colistin-resistant CRKp from blood cultures or other sites during the 30-day period when the initial blood culture was positive for colistin-susceptible CRKp.
Nephrotoxicity | 1 month
  Increase in serum creatinine to ≥1.5 times baseline which is known or presumed to have occurred within the prior 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Isler, MD, Principal Investigator — Sisli Hamidiye Etfal Training and Research Hospital; Önder Ergönül, MD, Study Director — Koç University
Locations (15):
- Turkey (Türkiye) (15):
  - Ankara University, Ankara
  - Başkent University, Ankara
  - Hacettepe University, Ankara
  - Ministry of Health, Ankara Training and Research Hospital, Ankara
  - Uluduağ University, Bursa
  - American Hospital, Istanbul
  - Cerrahpaşa University, Istanbul
  - Istanbul Bilim University, Istanbul
  - Istanbul Training and Research Hospital, Istanbul
  - İstanbul Sultan Abdülhamid Han Training and Research Hospital, Istanbul
  - Koç University, Istanbul
  - Marmara University, Istanbul
  - Ministry of Health Okmeydanı Training and Research Hospital, Istanbul
  - Ministry Of Health, Kartal Koşuyolu High Speciality Educational and Research Hospital, Istanbul
  - Dokuz Eylül University, Izmir

REFERENCES:
- [Background] Nordmann P, Naas T, Poirel L. Global spread of Carbapenemase-producing Enterobacteriaceae. Emerg Infect Dis. 2011 Oct;17(10):1791-8. doi: 10.3201/eid1710.110655. PMID 22000347
- [Background] Lee CR, Lee JH, Park KS, Kim YB, Jeong BC, Lee SH. Global Dissemination of Carbapenemase-Producing Klebsiella pneumoniae: Epidemiology, Genetic Context, Treatment Options, and Detection Methods. Front Microbiol. 2016 Jun 13;7:895. doi: 10.3389/fmicb.2016.00895. eCollection 2016. PMID 27379038
- [Background] Schwaber MJ, Carmeli Y. Carbapenem-resistant Enterobacteriaceae: a potential threat. JAMA. 2008 Dec 24;300(24):2911-3. doi: 10.1001/jama.2008.896. No abstract available. PMID 19109119
- [Background] Landman D, Georgescu C, Martin DA, Quale J. Polymyxins revisited. Clin Microbiol Rev. 2008 Jul;21(3):449-65. doi: 10.1128/CMR.00006-08. PMID 18625681
- [Background] Monaco M, Giani T, Raffone M, Arena F, Garcia-Fernandez A, Pollini S; Network EuSCAPE-Italy; Grundmann H, Pantosti A, Rossolini GM. Colistin resistance superimposed to endemic carbapenem-resistant Klebsiella pneumoniae: a rapidly evolving problem in Italy, November 2013 to April 2014. Euro Surveill. 2014 Oct 23;19(42):20939. doi: 10.2807/1560-7917.es2014.19.42.20939. PMID 25358041
- [Background] Hauck C, Cober E, Richter SS, Perez F, Salata RA, Kalayjian RC, Watkins RR, Scalera NM, Doi Y, Kaye KS, Evans S, Fowler VG Jr, Bonomo RA, van Duin D; Antibacterial Resistance Leadership Group. Spectrum of excess mortality due to carbapenem-resistant Klebsiella pneumoniae infections. Clin Microbiol Infect. 2016 Jun;22(6):513-9. doi: 10.1016/j.cmi.2016.01.023. Epub 2016 Feb 3. PMID 26850824
- [Background] Daikos GL, Tsaousi S, Tzouvelekis LS, Anyfantis I, Psichogiou M, Argyropoulou A, Stefanou I, Sypsa V, Miriagou V, Nepka M, Georgiadou S, Markogiannakis A, Goukos D, Skoutelis A. Carbapenemase-producing Klebsiella pneumoniae bloodstream infections: lowering mortality by antibiotic combination schemes and the role of carbapenems. Antimicrob Agents Chemother. 2014;58(4):2322-8. doi: 10.1128/AAC.02166-13. Epub 2014 Feb 10. PMID 24514083
- [Background] Tumbarello M, Viale P, Viscoli C, Trecarichi EM, Tumietto F, Marchese A, Spanu T, Ambretti S, Ginocchio F, Cristini F, Losito AR, Tedeschi S, Cauda R, Bassetti M. Predictors of mortality in bloodstream infections caused by Klebsiella pneumoniae carbapenemase-producing K. pneumoniae: importance of combination therapy. Clin Infect Dis. 2012 Oct;55(7):943-50. doi: 10.1093/cid/cis588. Epub 2012 Jul 2. PMID 22752516
- [Background] Rodriguez-Bano J, Gutierrez-Gutierrez B, Machuca I, Pascual A. Treatment of Infections Caused by Extended-Spectrum-Beta-Lactamase-, AmpC-, and Carbapenemase-Producing Enterobacteriaceae. Clin Microbiol Rev. 2018 Feb 14;31(2):e00079-17. doi: 10.1128/CMR.00079-17. Print 2018 Apr. PMID 29444952
- [Background] Paul M, Carmeli Y, Durante-Mangoni E, Mouton JW, Tacconelli E, Theuretzbacher U, Mussini C, Leibovici L. Combination therapy for carbapenem-resistant Gram-negative bacteria. J Antimicrob Chemother. 2014 Sep;69(9):2305-9. doi: 10.1093/jac/dku168. Epub 2014 May 28. PMID 24872346
- [Background] Zusman O, Altunin S, Koppel F, Dishon Benattar Y, Gedik H, Paul M. Polymyxin monotherapy or in combination against carbapenem-resistant bacteria: systematic review and meta-analysis. J Antimicrob Chemother. 2017 Jan;72(1):29-39. doi: 10.1093/jac/dkw377. Epub 2016 Sep 13. PMID 27624572
- [Background] Gutierrez-Gutierrez B, Salamanca E, de Cueto M, Hsueh PR, Viale P, Pano-Pardo JR, Venditti M, Tumbarello M, Daikos G, Canton R, Doi Y, Tuon FF, Karaiskos I, Perez-Nadales E, Schwaber MJ, Azap OK, Souli M, Roilides E, Pournaras S, Akova M, Perez F, Bermejo J, Oliver A, Almela M, Lowman W, Almirante B, Bonomo RA, Carmeli Y, Paterson DL, Pascual A, Rodriguez-Bano J; REIPI/ESGBIS/INCREMENT Investigators. Effect of appropriate combination therapy on mortality of patients with bloodstream infections due to carbapenemase-producing Enterobacteriaceae (INCREMENT): a retrospective cohort study. Lancet Infect Dis. 2017 Jul;17(7):726-734. doi: 10.1016/S1473-3099(17)30228-1. Epub 2017 Apr 22. PMID 28442293
- [Background] Falcone M, Russo A, Iacovelli A, Restuccia G, Ceccarelli G, Giordano A, Farcomeni A, Morelli A, Venditti M. Predictors of outcome in ICU patients with septic shock caused by Klebsiella pneumoniae carbapenemase-producing K. pneumoniae. Clin Microbiol Infect. 2016 May;22(5):444-50. doi: 10.1016/j.cmi.2016.01.016. Epub 2016 Feb 3. PMID 26850826
- [Background] Gonzalez-Padilla M, Torre-Cisneros J, Rivera-Espinar F, Pontes-Moreno A, Lopez-Cerero L, Pascual A, Natera C, Rodriguez M, Salcedo I, Rodriguez-Lopez F, Rivero A, Rodriguez-Bano J. Gentamicin therapy for sepsis due to carbapenem-resistant and colistin-resistant Klebsiella pneumoniae. J Antimicrob Chemother. 2015 Mar;70(3):905-13. doi: 10.1093/jac/dku432. Epub 2014 Oct 25. PMID 25344809
- [Background] Poirel L, Potron A, Nordmann P. OXA-48-like carbapenemases: the phantom menace. J Antimicrob Chemother. 2012 Jul;67(7):1597-606. doi: 10.1093/jac/dks121. Epub 2012 Apr 11. PMID 22499996
- [Background] Balkan II, Aygun G, Aydin S, Mutcali SI, Kara Z, Kuskucu M, Midilli K, Semen V, Aras S, Yemisen M, Mete B, Ozaras R, Saltoglu N, Tabak F, Ozturk R. Blood stream infections due to OXA-48-like carbapenemase-producing Enterobacteriaceae: treatment and survival. Int J Infect Dis. 2014 Sep;26:51-6. doi: 10.1016/j.ijid.2014.05.012. Epub 2014 Jul 3. PMID 24998423
- [Background] Navarro-San Francisco C, Mora-Rillo M, Romero-Gomez MP, Moreno-Ramos F, Rico-Nieto A, Ruiz-Carrascoso G, Gomez-Gil R, Arribas-Lopez JR, Mingorance J, Pano-Pardo JR. Bacteraemia due to OXA-48-carbapenemase-producing Enterobacteriaceae: a major clinical challenge. Clin Microbiol Infect. 2013 Feb;19(2):E72-9. doi: 10.1111/1469-0691.12091. Epub 2012 Dec 12. PMID 23231088
- [Background] Lowman W, Schleicher G. Antimicrobial treatment and outcomes of critically ill patients with OXA-48like carbapenemase-producing Enterobacteriaceae infections. Diagn Microbiol Infect Dis. 2015 Feb;81(2):138-40. doi: 10.1016/j.diagmicrobio.2014.09.023. Epub 2014 Oct 2. PMID 25497419
- [Background] Rojas LJ, Salim M, Cober E, Richter SS, Perez F, Salata RA, Kalayjian RC, Watkins RR, Marshall S, Rudin SD, Domitrovic TN, Hujer AM, Hujer KM, Doi Y, Kaye KS, Evans S, Fowler VG Jr, Bonomo RA, van Duin D; Antibacterial Resistance Leadership Group. Colistin Resistance in Carbapenem-Resistant Klebsiella pneumoniae: Laboratory Detection and Impact on Mortality. Clin Infect Dis. 2017 Mar 15;64(6):711-718. doi: 10.1093/cid/ciw805. PMID 27940944
- [Background] Machuca I, Gutierrez-Gutierrez B, Gracia-Ahufinger I, Rivera Espinar F, Cano A, Guzman-Puche J, Perez-Nadales E, Natera C, Rodriguez M, Leon R, Caston JJ, Rodriguez-Lopez F, Rodriguez-Bano J, Torre-Cisneros J. Mortality Associated with Bacteremia Due to Colistin-Resistant Klebsiella pneumoniae with High-Level Meropenem Resistance: Importance of Combination Therapy without Colistin and Carbapenems. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e00406-17. doi: 10.1128/AAC.00406-17. Print 2017 Aug. PMID 28559247
- [Background] Wright H, Bonomo RA, Paterson DL. New agents for the treatment of infections with Gram-negative bacteria: restoring the miracle or false dawn? Clin Microbiol Infect. 2017 Oct;23(10):704-712. doi: 10.1016/j.cmi.2017.09.001. Epub 2017 Sep 8. PMID 28893690
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338